CLINICAL TRIAL: NCT01705743
Title: Minimum Alveolar Concentration of Sevoflurane With 60% Nitrous Oxide Inducing Isoelectric EEG in Mid-aged Adults
Brief Title: Minimum Alveolar Concentration of Sevoflurane With Nitrous Oxide Inducing Isoelectric EEG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wei Mei, Associate Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TJMZK20120903
Record Dates: First submitted 2012-10-10; First posted 2012-10-12 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Middle Aged Patients; General Anesthesia
Keywords: anaesthesia; middle aged; minimal alveolar concentration; sevoflurane; nitrous oxide; isoelectric EEG
MeSH Terms: interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 Sevoflurane+Nitrous oxide (Active Comparator)
  Interventions: Drug: Sevoflurane+Nitrous oxide
- Group 2 Sevoflurane (Active Comparator)
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane+Nitrous oxide — 60% nitrous oxide +40% oxygen+ Sevoflurane
  Arms: Group 1 Sevoflurane+Nitrous oxide
Drug: Sevoflurane — 100% oxygen+ Sevoflurane
  Arms: Group 2 Sevoflurane

SUMMARY:
In order to investigate the effect of a combination effect of sevoflurane and nitrous oxide on cerebral electrical activity, the investigators determined the MAC of sevoflurane combined with nitrous oxide inducing isoelectric electroencephalogram (EEG) in 50% of the subjects (MACie) in middle aged subjects.

DETAILED DESCRIPTION:
Anaesthesia was induced by sevoflurane in oxygen. Cisatracurium 0.15 mg kg-1 was administered after loss of the lash reﬂex, then ventilated manually until the amplitude of T1 decreased to 0. Intubation was performed and switched to mechanical ventilation with a fresh gas flow of 2 L min-1. Anesthesia was maintained by sevoflurane or sevoflurane+60% nitrous oxide respectively. The surgical incision was performed at least 30 min after tracheal intubation, provided that the predetermined end-tidal sevoflurane concentration had been constant for at least 30 min and that the difference between inspired and end-tidal concentrations was less than 10%.

Brain electrical activity was measured using Narcotrend Monitor and S/5 Compact Anaesthesia Monitor, which displayed unprocessed EEG and burst suppression ratio, respectively. The design of the experiment is referred to the "Dixon up-and-down" method. To avid anaesthesia awareness, the first subject was designed to receive end-tidal sevoflurane concentration of 2.5 %. The presence or absence of isoelectric EEG (Entropy Module) of the preceding patient determined the end-tidal concentration of sevoflurane given to the next patient (with an increment size of 0.2%). The isoelectric EEG was considered as significant when the isoelectric state last for more than 1 min. The maximal burst suppression rate was recorded if isoelectric EEG was not reached.

ELIGIBILITY:
Inclusion Criteria:

* between 45 to 64 years old
* ASA physical status class 1 or 2
* elective abdominal surgery
* Informed Consent

Exclusion Criteria:

* history of neurological disease
* received central nervous system-active drugs
* cardiac ejection fraction less than 40%
* history of difficult intubation or anticipated difficult intubation
* daily alcohol consumption
* obesity, defined as a body-mass index of more than 30
* without informed consent
* others judged inappropriate as subjects for the study by the Study Chair

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
MACie | 30min
  Minimal Alveolar Concentration of sevoflurane and NO inducing isoelectric electroencephalogram (EEG) in 50% of the subjects (MACie)

CONTACTS AND LOCATIONS:
Overall Officials: Yuke Tian, MD., Study Chair — Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China